CLINICAL TRIAL: NCT01814605
Title: Ultrasound-guided Sciatic Nerve Block Using the Subgluteal Space Injection Approach: A Comparison With the Infragluteal Approach
Brief Title: Sciatic Nerve Block Using the Subgluteal Space Approach: A Comparison With the Infragluteal Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0060-A
Record Dates: First submitted 2013-02-11; First posted 2013-03-20 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Neuromuscular Blockade
Keywords: Sciatic Nerve Block; Subgluteal space; Infragluteal space

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subgluteal space group (Experimental): The patients in Subgluteal space group will receive sciatic block according to the approach described by Karmakar et al. Ultrasound scanning will be used to identify and mark the greater trochanter laterally and the ischial tuberosity medially. The midpoint will be designated with a marker and will be the site of needle entry.
  A 50 to 90 mm 22 G insulated needle will be inserted at the midpoint previously designated and advanced under real time guidance in an out-of-plane approach until the needle reaches the subgluteal space.
  Interventions: Procedure: Subgluteal space group
- Infragluteal space group (Active Comparator): The patients in this group will receive sciatic bock according to the approach described by Chan et al. Ultrasound scanning will be used to identify and mark the greater trochanter laterally and the ischial tuberosity medially. The midpoint between these two structures is a rough non-binding estimate of the approximate location of the sciatic nerve. After skin and transducer preparation, a curved 5 MHz(megahertz) transducer will be placed over the subgluteal region in a transverse plane to scan the sciatic nerve. A 50 to 90 mm 22 G needle is used and advanced under real time guidance in an out-of-plane approach until the needle tip is adjacent o the nerve.
  Interventions: Procedure: Infragluteal space group

INTERVENTIONS:
Procedure: Infragluteal space group — Sciatic Nerve Block "Infragluteal group": Ultrasound scanning will be used to identify and mark the greater trochanter laterally and the ischial tuberosity medially. The midpoint between these two structures is a rough non-binding estimate of the approximate location of the sciatic nerve. The sciatic nerve is usually found anterior (deep) to the gluteus maximus muscle and lateral to the origin of the biceps femoris muscle at the ischial tuberosity as well as medial to the greater trochanter.
  The end point of nerve block in this group is obtaining a circumferential local anesthetic spread around the sciatic nerve.
  Arms: Infragluteal space group
Procedure: Subgluteal space group — Subgluteal space group: The operator will identify the gluteus maximus and biceps femoris muscles at the level of the greater trochanter and ischial tuberosity and the infragluteal space.
  Arms: Subgluteal space group

SUMMARY:
A new ultrasound-guided "subgluteal space" approach to sciatic nerve block that has been recently described obviates the need to identify the sciatic nerve. The investigators hypothesize that the use of an ultrasound-guided subgluteal space injection to perform sciatic nerve block will increase the proportion of patients experiencing complete sensory block in both terminal branches of the Sciatic nerve in comparison to the same proportion in those who receive the block via ultrasound-guided infragluteal approach with circumferential injection in patients scheduled for unilateral TKA(total knee arthroplasty) surgeries.

DETAILED DESCRIPTION:
The subgluteal space technique is performed by injecting local anesthetics in the space sandwiched between the gluteus maximus and biceps femoris muscle at the level of the greater trochanter and ischial tuberosity rather than circumferentially around the nerve. The bone landmarks are particularly easier to identify because of the high acoustic mismatch and attenuation of bone. The end point of this technique is the distention of the subgluteal space to injection through the block needle. This new approach may translate in benefits including reducing block procedure time, reducing number of needle passes, reducing side effects (vascular complications), and ultimately block success.

The philosophy of injecting local anesthetics in designated anatomic spaces or between the fascial planes where nerves travel, as in the fascia iliaca block for example, is a time tested approach and has become more popular with the introduction of ultrasound because of the ease of visualizing fascia and bone in comparison to nerves under ultrasound. The call for injecting between planes and to stay away from nerves being blocked has found supporting evidence in trials involving ultrasound-guided brachial plexus block at the interscalene level.

One important potential advantage of the subgluteal space approach may be an increased safety margin created when distance is maintained between injecting needles and target nerves, an advantage that seems to make these injection techniques progressively more popular and to expand into a variety of single and continuous nerve blocks.

The investigators aim to compare the newly described ultrasound-guided subgluteal space block technique of the sciatic nerve to the currently practiced ultrasound-guided infragluteal sciatic nerve block with circumferential perineural spread in patients undergoing unilateral TKA surgery.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* ASA(American Society of Anesthesiologists physical status classification system) I-III patients undergoing unilateral TKA under spinal anesthesia and nerve blocks
* Ages 18-85
* BMI ≤ 38 Kg/m2

Exclusion Criteria:

* Chronic pain disorders
* Significant pre-existing neurological deficits or peripheral neuropathy affecting the lower extremity
* Abuse of drugs or alcohol
* Allergies to any medication included in the study protocol
* Contraindication to spinal anesthesia
* History of significant psychiatric conditions that may affect patient assessment
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Complete sensory block in the distribution of both terminal branches of the sciatic nerve. | up to 30 minutes
  The independent observer, blinded to the block technique used, will assess patients for sensory and motor block every 5 minutes for 30 minutes or until start of surgery

SECONDARY OUTCOMES:
Block procedure time | until local anesthetic injection has been completed
  The time elapsed from ultrasound probe positioning until local anesthetic injection has been completed

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Allen HW, Liu SS, Ware PD, Nairn CS, Owens BD. Peripheral nerve blocks improve analgesia after total knee replacement surgery. Anesth Analg. 1998 Jul;87(1):93-7. doi: 10.1097/00000539-199807000-00020. PMID 9661553
- [Background] Cook P, Stevens J, Gaudron C. Comparing the effects of femoral nerve block versus femoral and sciatic nerve block on pain and opiate consumption after total knee arthroplasty. J Arthroplasty. 2003 Aug;18(5):583-6. doi: 10.1016/s0883-5403(03)00198-0. PMID 12934209
- [Background] Weber A, Fournier R, Van Gessel E, Gamulin Z. Sciatic nerve block and the improvement of femoral nerve block analgesia after total knee replacement. Eur J Anaesthesiol. 2002 Nov;19(11):834-6. doi: 10.1017/s0265021502221353. No abstract available. PMID 12442936
- [Derived] Abdallah FW, Chan VW, Koshkin A, Abbas S, Brull R. Ultrasound-guided sciatic nerve block in overweight and obese patients: a randomized comparison of performance time between the infragluteal and subgluteal space techniques. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):547-52. doi: 10.1097/AAP.0000000000000016. PMID 24121610